CLINICAL TRIAL: NCT05256927
Title: Is Milk Associated with Glycemia in the NICU (MAGIC) a Study in the NICU
Brief Title: Is Milk Associated with Glycemia in the NICU
Acronym: MAGIC
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Bridget Young, Assistant Professor, University of Rochester
Other Study IDs: STUDY00006851; 1R03DK131219 (NIH)
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All Participants

SUMMARY:
The purpose of this study is to determine if concentrations of hormones in prepared human milk (HM) feeds are associated with metabolic disturbances in the recipient premature infant. To do so, prospectively 100 infants receiving HM-derived fortifiers as part of clinical care will be studied, saving aliquots of daily prepared feeds until any fortification ceases.

DETAILED DESCRIPTION:
The purpose of this study is to determine if concentrations of these hormones in prepared HM feeds are associated with metabolic disturbances in the recipient infant. A prospectively study 100 infants receiving HM-derived fortifiers as part of clinical care, saving aliquots of daily prepared feeds until any fortification ceases. Insulin and PTHrP will be compared in feeds from matched days when metabolic disturbances were documented vs not; each infant serving as a control.

Hypothesis 1 Feed dose of insulin and PTHrP will be higher from days when hypoglycemia and hypercalcemia are observed, respectively, vs control days when metabolic disturbances are not observed.

Hypothesis 2: Over time, daily feed dose of insulin will correlate with average daily blood glucose in infants receiving HM products.

ELIGIBILITY:
Inclusion Criteria:

* Infants eligible to receive human milk (HM)-derived fortifiers. To qualify for these fortifiers, infants must be born <30 weeks gestation and/or weigh <1250g at birth. Enteral or oral feeding modes both qualify for participation. Additional supplementation to feeds beyond HM-derived fortifier (such as medium-chain triglycerides) is acceptable.
* Infants initially on intravenous nutrition will still be eligible for consent. Feed sample collections from these infants will commence once they advance to consume HM-based feeds once HM-derived fortifier is prescribed.

Exclusion Criteria:

* Infants diagnosed with congenital disorders that impact glucose or calcium metabolism will be excluded.
* Infants with conditions necessitating specialized diets (ex: chylothorax) will also be excluded.
* Non-English speaking subjects will be excluded as the team of study personnel includes those that speak English only.

Ages: 0 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants admitted to the University of Rochester Medical Center that are <30 weeks gestation and/or weigh <1250g at birth.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Insulin concentration in prepared feeds | 3 months
  We will measure final insulin concentrations in enteral feed preparations that contain some portion of human milk.
Parathyroid hormone related protein (PTHrP) concentration in prepared feeds | 3 months
  We will measure final PTHrP concentrations in enteral feed preparations that contain some portion of human milk.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No